CLINICAL TRIAL: NCT03804541
Title: A Single-center, Open-label, Single-dose Phase I Study to Investigate the Absorption, Metabolism and Excretion of [14C]Ensartinib (X-396) After a Single Oral 200mg (100µCi) Dose in Healthy Chinese Male Subjects
Brief Title: The Absorption, Metabolism and Excretion of [14C]Ensartinib in Human
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTP-44316
Record Dates: First submitted 2018-12-26; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: ALK-POSITIVE NSCLC
MeSH Terms: interventions — ensartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]Ensartinib (Experimental): To investigate the absorption properties, as well as to evaluate the mass balance and elucidate the pathways of biotransformation after a single oral dose (200mg, 100µCi) of [14C]Ensartinib to healthy Chinese male subjects。
  Interventions: Drug: Ensartinib

INTERVENTIONS:
Drug: Ensartinib — A novel, potent ALK inhibitor.The ALK inhibitor ensartinib has been validated in potency and selectivity assays indicating that it is more selective and up to 10 times more potent than competitive ALK inhibitors. Ensartinib has been active in animal models of non-small cell lung cancer (NSCLC) and neuroblastoma, a childhood cancer. Importantly, ensartinib has shown activity in models with ALK mutations that confer resistance to other small molecule ALK inhibitors.
  Other Names: X-396

SUMMARY:
This is a single-center, open-label, single-dose phase I study to investigate the absorption, metabolism and excretion of [14C] Ensartinib in healthy Chinese male subjects. The study will be conducted into two steps：Firstly, 2 subjects are enrolled in to participate in the pilot study to grope for the completion date of plasma, urine and feces sampling on the 3rd day post-dose and onwards. Then, the collection time of blood and excreta samples (urine and feces) from the subsequent 4-6 subjects will be adjusted according to the pilot study.

DETAILED DESCRIPTION:
Subjects who had signed informed consent and meet inclusion criteria and no exclusion criteria are admitted to Phase I Clinical Unit two days prior to dosing (D-2). On the morning of Day 1 before dosing, subjects will be transferred to nuclear medical ward. And after an overnight fast of at least 10 h, subjects will receive a single oral dose of 200 mg (100 μCi) of [14C]Ensartinib as an oral suspension. Then, after two days of the dosing, subjects will be transferred back to Phase I Clinical Unit ward and confined to this unit until blood or excreta sampling and safety monitoring at the designated time points or intervals are complete

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for study participation if he meets the following criteria:

1. healthy male volunteers between the ages of 18 to 50 years old, inclusive;
2. Body weight >=50 kg, Body mass index (body weight(kg)/hight2(m2)) between 19 and 26 kg/m2 (inclusive);
3. Normal physical findings, clinical laboratory values, vital signs and 12-lead ECG, or any abnormality that is non-clinically significant;
4. Male subjects of reproductive potential with partners will be instructed to, and must be willing to practice a highly effective method of birth control for the duration of the study and continuing 1 year after discontinuing treatment with the investigational product. Highly effective methods of birth control include using condom, contraceptive sponge, contraceptive gel, contraceptive film, intrauterine device, oral or injectable contraceptive pill, hypodermic implants or others;
5. Must understand, and voluntarily sign the informed consent, comply with the requirements of the study

Exclusion Criteria:

A subject will not be eligible for study participation if he meets any of the exclusion criteria:

1. History of or current clinically significant cardio, pulmonary, endocrine, metabolism, renal, hepatic, gastrointestinal, dermatology, infection, hematology, neurological, mental disease or disorder;
2. Positive test for HBsAg, HBeAg, anti-HCV, anti-HIV or syphilis antibody;
3. History of clinically significant disease or infection within 1 month before entering the study;
4. Abnormality in blood pressure, including hypertensive BP (SBP>=140 mmHg, or DBP >=90 mmHg), or hypotensive BP(SBP<90 mmHg, or DBP <=55 mmHg), Pulse rate<55 bpm or >100 bpm;
5. Long-QT syndrome or family history of it, or QTcB interval > 450 ms; intraventricular blocks or left/right bundle branch block or QRS>120ms; frequent ventricular ectopic beats (any 10s ECG ventricular premature beat >= 1 in screening period); or abnormal resting heart rate (> 100 bpm)
6. The following abnormal clinical laboratory values

   1. HGB < LLN, and is judged as clinically significant by the investigator；
   2. Abnormal ALP, ALB,TP,CRE,ALT,AST,BIL,BUN, GLU value, and is judged as clinically significant by the investigator;
7. Received any drug within 14 days before taking the investigational drug, including any prescription drug, OTC drug or herbal drug, except for vitamins and paracetamol;
8. History of or current swallowing disorder, active gastrointestinal diseases, or other diseases that significantly affect absorption, distribution, metabolism and excretion of drugs;
9. Chronic constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease;
10. Hemorrhoids or perianal disease with regular/perianal bleeding;
11. Allergies, have allergies to two or more drugs or foods; or have known allergies to the components of the drug (microcrystalline cellulose, stearic acid, hydroxypropyl methylcellulose);
12. Have donated 500ml or more of blood or plasma 2 months prior to the study drug administration, or more than 50ml within 2 weeks prior to administration;
13. Vaccination was administered within 6 months prior to screening or during screening;
14. History of drug or alcohol abuse;
15. Smoking (> 10 cigarette / day), drinking (> 15 g, pure alcohol / day, equivalent to 450 ml beer, 150 ml wine or 50 ml low-alcohol liquor), or abusing drugs(MOP, METmAMP, MTD, THC, AMP positive) within last 3 months;
16. Subject with mentally ill and could not understand the property, scope and possible consequences of the study;
17. subject in prison or whose freedom is restricted by administrative or legal issues;
18. Failure to comply with clinical study protocols, such as non-cooperation, follow-up visit and completion of entire study;
19. Investigator, pharmacist, CRC or research associate;
20. Investigators think that subjects are not suitable to participate in the study;
21. Subjects who have participated in radiolabeled clinical study prior to drug administration;
22. Significant radiation exposure within one year prior to drug administration (more than one exposure from chest X-ray, CT scan, or barium meal examination and radiation-related occupations).

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2018-12-28 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Radioactivity concentration of each plasma sample | Day1-Day15
  Use liquid scintillation counter to evaluate Radioactivity concentration of each plasma（DPM/ml) sample
Radioactivity concentration of each urine samples | Day1-Day15
  Use liquid scintillation counter to evaluate Radioactivity concentration of each urine（DPM/ml） sample
Radioactivity concentration of each feces sample | Day1-Day15
  Use liquid scintillation counter to evaluate Radioactivity concentration of each feces（DPM/g） sample
Total recovery of radioactivity in urine and feces | Day1-Day15
  Calculate the total radioactivity in urine and feces based on the radioactivity concentration of each sample.

SECONDARY OUTCOMES:
Plasma drug concentrations | Day1-Day15
  To determine the plasma concentrations of Ensartinib with validated LC-MS/MS method for obtaining its pharmacokinetics parameters;
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | Day1-Day15
  According to CTCAE v4.03, the number and frequency of adverse events after a single dose of test drug were assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shao, Principal Investigator — Jiangsu Province Hospital Affiliated to Nanjing Madical University of Medicine
Locations (1):
- Jiangsu Province Hospital Affiliated to Nanjing Madical University of Medicine, Nanjing, Jiangsu Provence, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nijenhuis CM, Schellens JH, Beijnen JH. Regulatory aspects of human radiolabeled mass balance studies in oncology: concise review. Drug Metab Rev. 2016 May;48(2):266-80. doi: 10.1080/03602532.2016.1181081. Epub 2016 May 17. PMID 27186889
- [Background] Penner N, Klunk LJ, Prakash C. Human radiolabeled mass balance studies: objectives, utilities and limitations. Biopharm Drug Dispos. 2009 May;30(4):185-203. doi: 10.1002/bdd.661. PMID 19544285
- [Derived] Zhou S, Liu W, Zhou C, Zhang L, Xie L, Xu Z, Wang L, Zhao Y, Guo L, Chen J, Ding L, Mao L, Tao Y, Zhang C, Ding S, Shao F. Mass balance, metabolic disposition, and pharmacokinetics of [14C]ensartinib, a novel potent anaplastic lymphoma kinase (ALK) inhibitor, in healthy subjects following oral administration. Cancer Chemother Pharmacol. 2020 Dec;86(6):719-730. doi: 10.1007/s00280-020-04159-0. Epub 2020 Oct 12. PMID 33044566
- See also: [6] CFR 361.1 Radioactive Drugs for Certain Research Uses. — http://edocket.access.gpo.gov/cfr_2008/aprqtr/pdf/21cfr36.